CLINICAL TRIAL: NCT01701687
Title: The Feasibility of Liver Biomarkers as Prognostic Markers in Decompensated Alcoholic Liver Disease
Brief Title: Biomarkers for the Prognosis of Decompensated Alcoholic Liver Disease
Acronym: BANDED
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 12050
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Alcoholic Liver Diseases; Decompensated Cirrhosis
Keywords: Cirrhosis; Alcoholic liver disease; Decompensated liver cirrhosis; Hazardous alcohol
MeSH Terms: conditions — Liver Diseases, Alcoholic; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and urine stored at -80 degrees centigrade under written patient consent
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Decompensated Alcoholic Cirrhosis: Recruited patients will have diagnosed liver cirrhosis (histological, radiological or accepted clinical parameters)admitted with an episode of decompensation. Patients must still be drinking hazardous alcohol quantities (>14 units for women, >21 units for men) at study enrollment

SUMMARY:
Fibroscan is a non invasive imaging investigation which measures liver stiffness, known to correlate well with liver scarring and cirrhosis on liver biopsy. Indocyanine green is an inert dye which is purely extracted from the blood by liver cells, and is hence an excellent marker of both liver cell function and overall liver blood flow. There is little data for either of these biomarkers regarding outcomes in alcoholic liver disease. We aim to establish the accuracy of these liver biomarkers in predicting important liver related outcomes (death, transplantation and hospital readmission with cirrhosis related consequences) in patients with severe (decompensated) alcoholic liver disease. Moreover, we will assess whether the serial measurement of biomarkers has any impact on alcohol abstinence, motivation or quality of life. Over an 18 month period, 125 consecutive hospital inpatients with decompensated alcoholic liver disease will undergo baseline biomarker measurement, routine blood and urine tests and qualitative questionnaires. These will be measured during their initial hospital admission (0 months) with subsequent repeat measurement during follow up visits at 1, 2, 4 and 6 months. Each study visit time will be in the region of 30-40 minutes to complete these investigations. The end of the study for individual patients will be patient death, liver transplantation or 6 month from study enrolment; whichever occurs first.

DETAILED DESCRIPTION:
This is a single centre longitudinal cohort feasibility pilot study of patients with decompensated alcoholic liver disease. We aim to recruit 125 consecutive patients with decompensated alcoholic liver disease over an 18 month period. This number is based upon approximately 10 admissions per month to acute liver services with decompensated alcoholic liver disease and includes a presumed 20% dropout rate during follow up, giving a total cohort of 100 patients. Patients will undergo a maximum of 6 months follow up following study recruitment.

The purposes of this study are:

1. To assess the performance of diagnostic liver biomarkers (Indocyanine Green, Fibroscan and blood and urinary biomarkers) in predicting mortality in decompensated alcoholic liver disease.
2. To compare the diagnostic and prognostic end points of these biomarkers with existing cirrhosis prognostic scoring systems (Child Pugh, MELD and UKELD).
3. To assess the performance of diagnostic biomarkers as a therapeutic aid to quality of life and alcohol abstinence.

Potentially eligible patients i.e. adults with decompensated liver disease with alcohol as a major co-factor, and acutely admitted secondary to sequelae of hepatic decompensation, will be approached by an existing member of their clinical care team (The CI & Co-Investigators form part of this team). Any patient who decides to take part in the study will have a baseline inpatient study visit either on their inpatient ward or to the NDDC Biomedical Research Unit (BRU). Subsequent follow up visits will be to the BRU.

Inclusion Criteria:

* Male or female patients 18-75 years of age
* Diagnosis of cirrhosis based upon:

  * a) Histological confirmation
  * b) Combination of clinical and radiological criteria
  * c) Validated non invasive biomarker
* Alcohol as the primary aetiology for liver cirrhosis
* Hospital admission related to decompensated liver disease (e.g. ascites, varices, sepsis, alcoholic hepatitis)
* Active alcohol drinking prior to index hospital admission

Exclusion Criteria:

* Grade 3 or 4 hepatic encephalopathy
* Hepatocellular carcinoma
* Active non hepatic malignancy
* Known complete portal vein thrombosis
* Alcohol abstinence at time of index hospital admission
* Pregnancy
* Active cardiac devices

The research visit will require measurement of ICG clearance, Fibroscan, blood tests, urine tests and questionnaires. They will then be required to attend study visits at 1, 2, 4 and 6 months following the baseline study visit, after which study follow up will cease.

Patients will undergo study visits at the following intervals:

* Baseline visit (study visit 0)
* 1 month (study visit 1)
* 2 months (study visit 2)
* 4 months (study visit 3)
* 6 months (study visit 4)

The following data will be collected for the purposes of this research project at the baseline and subsequent study visits:

* Collection of demography, anthropometry, drug history, smoking, alcohol intake, blood pressure, full blood count, renal function, liver function, coagulation and serum samples
* Brief abdominal examination to detect presence of moderate to severe ascites (for the purposes of Child Pugh score measurement)
* ICG analysis
* Transient elastography (Fibroscan)
* Blood and urinary biomarkers (proteomics and metabonomics)
* Chronic Liver Disease Quality of Life Questionnaire
* Alcohol intake assessments (28 Day AUDIT tool)
* Alcohol STAR tool for qualitative assessment (to assess the influence of Fibroscan/ICG readings on motivation, beliefs and alcohol abstinence)

Demography and history are taken as part of normal clinical care. All patients will be offered standard follow up from both outpatient hepatology clinic and hospital alcohol liaison services throughout the period of study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18-75 years of age
* Diagnosis of cirrhosis based upon:

  * a) Histological confirmation
  * b) Combination of clinical and radiological criteria
  * c) Validated non invasive biomarker
* Alcohol as the primary aetiology for liver cirrhosis
* Hospital admission related to decompensated liver disease (e.g. ascites, varices, sepsis, alcoholic hepatitis)
* Active alcohol drinking prior to index hospital admission

Exclusion Criteria:

* Grade 3 or 4 hepatic encephalopathy
* Hepatocellular carcinoma
* Active non hepatic malignancy
* Known complete portal vein thrombosis
* Alcohol abstinence at time of index hospital admission
* Pregnancy
* Active cardiac devices (e.g. cardiac pacemaker, implantable cardioverter defibrillator)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentially eligible patients are adult patients with decompensated liver disease with alcohol as a major co-factor, and acutely admitted secondary to sequelae of hepatic decompensation. 100 patients will be recruited for baseline visit over an 30 month study enrolment period, with a 6 month follow up period for all patients.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Liver Related Death | 6 months
  The proportion of deaths up to 6 months from the baseline visit directly attributable to consequences of cirrhosis

SECONDARY OUTCOMES:
Non-Liver related death | 6 months
  Mortality unrelated to liver disease up to 6 months from baseline study visit
Hospital Readmission | 6 months
  Hospital readmission secondary to complications of cirrhosis
Alcohol abstinence | 6 months
  Proportion of patients abstinent from alcohol at the 6 month timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Neil Guha, MRCP, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Notts, United Kingdom